CLINICAL TRIAL: NCT03824795
Title: An Exploratory, Open Labelled, Phase IIa Study to Assess Safety, Tolerability and Efficacy of Incremental Doses of MGB-BP-3 in Patients With Clostridium Difficile-associated Diarrhea (CDAD)
Brief Title: Study to Assess Safety, Tolerability and Efficacy of Incremental Doses of MGB-BP-3 in Patients With CDAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MGB Biopharma Limited (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1011464; 2015-000489-73 (EudraCT Number); 129507 (Other: FDA IND Number); MGB-BP-3-201 (Other: Syneos Health Protocol Number)
Record Dates: First submitted 2019-01-24; First posted 2019-01-31 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; CDAD; MGB-BP-3; Novel anti-infective; Efficacy; Tolerability; Safety; Phase IIa
MeSH Terms: conditions — Clostridium Infections | interventions — MGB-BP-3

STUDY DESIGN:
Intervention Model Description: This is an open-label study with 3 sequential groups of 10 patients with CDAD with a staggered start.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: 125mg b.i.d. for 10 days (Active Comparator): Patients will be administered an oral dose of 125mg b.i.d. MGB-BP-3 for 10 days (Day 1 to Day 10).
  Interventions: Drug: MGB-BP-3
- Group 2: 250mg b.i.d. for 10 days (Active Comparator): Patients will be administered an oral dose of 250mg b.i.d. MGB-BP-3 for 10 days (Day 1 to Day 10).
  Interventions: Drug: MGB-BP-3
- Group 3: 500mg b.i.d. for 10 days (Active Comparator): Patients will be administered an oral dose of 500mg b.i.d. MGB-BP-3 for 10 days (Day 1 to Day 10).
  Interventions: Drug: MGB-BP-3

INTERVENTIONS:
Drug: MGB-BP-3 — MGB-BP-3
  Other Names: No other names - not applicable

SUMMARY:
The objective of this Phase IIa study is to assess the safety, tolerability, and efficacy of incremental doses of MGB-BP-3 in patients with Clostridium difficile-associated diarrhea (CDAD).

DETAILED DESCRIPTION:
This is an exploratory, Phase IIa, open-label study assessing the safety, tolerability, and efficacy of incremental doses of MGB-BP-3 with 3 sequential groups of 10 patients with CDAD. Patients will be administered an oral dose of MGB-BP-3 for 10 days (Day 1 to Day 10). At the end of the treatment period, patients will be followed for up to 8 weeks to assess the incidence of disease recurrence.

ELIGIBILITY:
Main Inclusion Criteria:

1. Age 18 years or older of any gender.
2. Inpatients and/or outpatients who are able to attend all scheduled visits.
3. Patients with the first episode or the first recurrence of mild or moderate CDAD.
4. Confirmed diagnosis of mild or moderate CDAD as defined by the Infectious Diseases Society of America/Society for Healthcare Epidemiology of America guidelines.

Main Exclusion Criteria:

1. Patients with severe complicated CDAD (including hypotension or shock, ileus, megacolon, pseudomembranous colitis).
2. A white blood cell count higher than 15,000 cells/mL.
3. A serum creatinine level greater than or equal to 1.5 times ULN.
4. Elevated liver enzymes alanine aminotransferase and aspartate aminotransferase greater than ULN.
5. Inflammatory bowel disease (ulcerative colitis or Crohn's disease), microscopic colitis, or irritable bowel syndrome with chronic diarrhea.
6. Any other non-C difficile diarrhea.
7. Received treatment with a fecal transplant within 7 days and/or is anticipated to receive a fecal transplant during the study.
8. Major gastrointestinal surgery (ie, significant bowel resection) within 3 months of enrollment (does not include appendectomy or cholecystectomy).
9. Received laxatives within the previous 48 hours.
10. Pregnant or lactating women.
11. Prior (within 180 days of Screening) or current use of anti-toxin antibodies.
12. Have received a vaccine against C difficile.
13. Any condition for which, in the opinion of the investigator, the treatment may pose a health risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-04-03 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by the Investigator, as per CTCAE v.5.0. | 40 days
  Incidence of treatment emergent adverse events (Safety and Tolerability of up to 3 incremental doses of MGB-BP-3 in patients with CDAD).
Initial cure rate at 12 days post initiation of therapy. | 12 days
  Initial clinical cure is defined as resolution of diarrhea (<3 bowel movements with unformed stools within 24 hours [Type 5, 6, or 7 bowel movement on the Bristol Stool Chart] for patients for 2 consecutive days), maintained for the subsequent duration of therapy (1 day of exacerbation and then return to the resolved state is acceptable), with no further requirement for CDAD therapy, assessed by EOT and sustained for 2 days after the end of the 10-day initial treatment course.

SECONDARY OUTCOMES:
CDAD Recurrence | Up to 8 weeks
  Recurrence of CDAD within 4 weeks (8 weeks optional) post end of treatment.
Peak plasma concentration (Cmax). | 10 days
  Days 1, 5 and 10.
Time to peak plasma concentration (Tmax). | 10 days
  Days 1, 5 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Ravic, MD, Study Director — MGB Biopharma Ltd.
Locations (9):
- United States (8):
  - Florida International Medical Research, Miami, Florida
  - Omega Research Maitland LLC, Orlando, Florida
  - Snake River Research PLLC, Idaho Falls, Idaho
  - Ochsner Clinic Foundation Infectious Disease Research, New Orleans, Louisiana
  - Anne Arundel Medical Centre, Annapolis, Maryland
  - Mercury Street Medical Group PLLC, Butte, Montana
  - Biopharma Informatic LLC, Houston, Texas
  - Verity Research Inc., Fairfax, Virginia
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No